CLINICAL TRIAL: NCT00962923
Title: Allogeneic Mesenchymal Stem Cells Transplantation for Systemic Sclerosis (SSc)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJGLYY003
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Systemic Sclerosis; Mesenchymal Stem Cells
Keywords: Systemic sclerosis; Mesenchymal Stem Cells; Transplantation
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Stem Cells (AlloMSC) — Allogeneic mesenchymal stem cells will be infused intravenously (single dose, 10^6 cells/kg body weight).

SUMMARY:
This study will explore safety and efficacy of allogeneic mesenchymal stem cells transplantation (MSCT) to treat patients with diagnosis of systemic sclerosis(SSc) who have been resistant to multiple standard treatments. The underlying hypothesis is that the SSc condition is caused by an abnormal immune homeostasis that can be restored by MSCT.

DETAILED DESCRIPTION:
* To test a new approach using allogeneic derived mesenchymal stem cell based therapy (MSCT) to treat refractory SSc
* To determine the disease-free survival in SSc patients treated with MSCT
* To assess adverse events of allogeneic MSC transplantation
* To assess the association of remission for organ function, clinical score and SSc serology levels at baseline with disease-free survival

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the American College of Rheumatology (former American Rheumatism Association - ARA) for SSc
* Rapidly progressive disease <2 years duration with a modified Rodnan skin score(mRSS) above 20, plus ESR >25 mm/first h and/or Hb <11 g/dL, not explained by other causes than active SSc
* lung involvement: with a vital capacity (VC) or DLCO below 70% predicted, or a mean pulmonary artery pressure (PAP) above 40 mmHg (measured by echocardiography)
* digestive tract involvement: with serum albumin ,25 g/L or weight loss exceeding 10% body weight in the preceding year
* kidney involvement: with 24-h urinary protein above 0.5 g or serum creatinine above 120 mmol/L

Exclusion Criteria:

* Uncontrolled arrhythmia, echocardiographic left ventricular ejection fraction (LVEF) <50% or mean PAP >50 mmHg, DLCO<45% of predicted
* Creatinine clearance <20 ml/min
* Platelets<80 000/mm3, haemorrhagic cystitis
* (4) HIV or HTLV1 seropositivity, malignancy, pregnancy, a cardiac or vascular prosthesis, and no vascular access

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
mRSS score,HRQOL score, SF-36 score for SSc patients | monthly

SECONDARY OUTCOMES:
Remission for organ function, VC, DLCO, PAP, serum albumin, serum creatitin, weight loss, 24h proteinuria | every three month
SSc Serology(ATA,ACA,ANA,anti-ssDNA,anti-dsDNA,IgM,IgG,and IgA,complement C3 and C4 | every three month
Change of peripheral blood B and T cells | every three month

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Sun L, Akiyama K, Zhang H, Yamaza T, Hou Y, Zhao S, Xu T, Le A, Shi S. Mesenchymal stem cell transplantation reverses multiorgan dysfunction in systemic lupus erythematosus mice and humans. Stem Cells. 2009 Jun;27(6):1421-32. doi: 10.1002/stem.68. PMID 19489103
- [Background] Liang J, Zhang H, Hua B, Wang H, Wang J, Han Z, Sun L. Allogeneic mesenchymal stem cells transplantation in treatment of multiple sclerosis. Mult Scler. 2009 May;15(5):644-6. doi: 10.1177/1352458509104590. PMID 19389752
- [Background] Zhou K, Zhang H, Jin O, Feng X, Yao G, Hou Y, Sun L. Transplantation of human bone marrow mesenchymal stem cell ameliorates the autoimmune pathogenesis in MRL/lpr mice. Cell Mol Immunol. 2008 Dec;5(6):417-24. doi: 10.1038/cmi.2008.52. PMID 19118507
- [Background] Sun LY, Zhang HY, Feng XB, Hou YY, Lu LW, Fan LM. Abnormality of bone marrow-derived mesenchymal stem cells in patients with systemic lupus erythematosus. Lupus. 2007;16(2):121-8. doi: 10.1177/0961203306075793. PMID 17402368
- [Derived] Alip M, Wang D, Zhao S, Li S, Zhang D, Duan X, Wang S, Hua B, Wang H, Zhang H, Feng X, Sun L. Umbilical cord mesenchymal stem cells transplantation in patients with systemic sclerosis: a 5-year follow-up study. Clin Rheumatol. 2024 Mar;43(3):1073-1082. doi: 10.1007/s10067-024-06865-z. Epub 2024 Jan 11. PMID 38206544
- [Derived] Zhang H, Liang J, Tang X, Wang D, Feng X, Wang F, Hua B, Wang H, Sun L. Sustained benefit from combined plasmapheresis and allogeneic mesenchymal stem cells transplantation therapy in systemic sclerosis. Arthritis Res Ther. 2017 Jul 19;19(1):165. doi: 10.1186/s13075-017-1373-2. PMID 28724445
- [Derived] Akiyama K, Chen C, Wang D, Xu X, Qu C, Yamaza T, Cai T, Chen W, Sun L, Shi S. Mesenchymal-stem-cell-induced immunoregulation involves FAS-ligand-/FAS-mediated T cell apoptosis. Cell Stem Cell. 2012 May 4;10(5):544-55. doi: 10.1016/j.stem.2012.03.007. Epub 2012 Apr 26. PMID 22542159